CLINICAL TRIAL: NCT06300749
Title: The Effect of Chiropractic Cervical Manipulation on Pain, Functionality and Grip Strength in Patients With Lateral Epicondylitis
Brief Title: Effectiveness of Chiropractic Cervical Manipulation in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesut Arslan (Other)
Responsible Party: Sponsor-Investigator, Mesut Arslan, Assistant Professor, Bitlis Eren University
Organization: Bitlis Eren University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LE-CCM
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Chiropractic Cervical Manipulation
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chiropractic Cervical Manipulation Group (CCMG) (Experimental): Patients in both groups were placed in supine position and manipulation was applied to patients in the chiropractic cervical manipulation group.
  Interventions: Other: Chiropractic Cervical Manipulation
- Control Group (CG) (Sham Comparator): Patients in both groups were placed in supine position and manipulation was applied to patients in the chiropractic cervical manipulation group.
  Interventions: Other: Sham Technique Practice

INTERVENTIONS:
Other: Chiropractic Cervical Manipulation — In the chiropractic cervical manipulation group, the patient was placed in the supine position. The therapist moved to the patient's head, identified the C5-C6 segment by palpation, and manually performed spinal manipulation from the right side using the "cervical rotary break/index push" technique since the dominant side of the patients was the right extremity. In the cervical rotary break/index thrust technique, the lateral aspect of the practitioner's index finger was placed in contact with the posterior aspect of the participant's C5 facet joint, and a rotational thrust was performed between the C5-C6 vertebrae.
  Arms: Chiropractic Cervical Manipulation Group (CCMG)
Other: Sham Technique Practice — The sham technique can be defined as a technique that does not have any therapeutic effect and is preferred to determine whether the efficacy of another technique is superior. The patient was placed in the supine position. The therapist moved to the patient's head, and the C5-C6 segment localized in the lower cervical region was detected by palpation. The C5-C6 segment was positioned to perform chiropractic cervical manipulation and waited for 30 seconds without any pushing force.
  Arms: Control Group (CG)

SUMMARY:
İt is aimed to examine the effect of chiropractic cervical manipulation on pain, functionality and grip strength in patients with lateral epicondylitis and whether it is preferable to placebo.

DETAILED DESCRIPTION:
Lateral Epicondylitis (LE) is known as chronic symptomatic degeneration of the forearm common extensor tendon attachment at the humeral ectochondyle. It is one of the most common overuse syndromes today and is characterized by loss of function and pain due to an inflammatory reaction that occurs during stretching of the condyle.

The main goals of the treatments are to relieve pain, reduce overload on the arm and elbow joints, accelerate the healing process and enable the patient to regain functionality in daily life activities at the optimum time. Many treatment methods have been applied for this purpose, and the number of studies on the effectiveness of manual applications is increasing. Among manual applications, chiropractic applications have recently attracted attention.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 20-50 years,
* (2) dominant right extremity and ipsilateral lateral epicondylitis,
* (3) full range of motion in the cervical region,

Exclusion Criteria:

* (1) spinal root compression (radiculopathy),
* (2) neurologic symptoms such as loss of strength in the lower extremities, upper extremities and face, numbness, involuntary movements, abnormal gait pattern, dizziness, nausea/vomiting of unknown cause, swallowing and speech difficulties,
* (3) pregnancy,
* (4) presence of active malignancies,
* (5) positive pre- manipulative vertebrobasilar insufficiency test,
* (6) use of anticoagulant and antiaggregant drugs,
* (7) history of previous cervical surgery or whiplash,
* (8) acute inflammatory disease,
* (9) positive results of the test performed before manipulation in the cervical spine (foraminal compression test,
* (10) any deformity in the New York Posture analysis,
* (11) unwillingness to participates

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale (NPS) | Pain was evaluated immediately before and immediately after the application.
  The patient is asked to indicate the value of their pain on the scale. During the assessment, an 11-point scale is used, with "0" representing "no pain" and "10" meaning "the most severe pain imaginable".
Grip Strength | Grip Strength parameter was evaluated immediately before and immediately after the application.
  Consistent with the American Hand Therapy Association's hand grip dynamometer recommendations and previous research, participants sat in a chair with the device in the dominant hand, wrists in a neutral position and elbows bent at a 90° angle. Three repeated measurements were taken, and averages were calculated.
Patient Rated Tennis Elbow Evaluation (PRTEE) | PRTEE parameter was evaluated immediately before and immediately after the application.
  A 15-item questionnaire was used to evaluate pain and disability. The questionnaire includes three subscales, with each item scored from 0 to 10. The total score ranges from 0 to 100, where higher scores indicate more pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No